CLINICAL TRIAL: NCT03885271
Title: Outcomes of the Hall Technique and Conventional Pulp Therapy for the Management of Caries in Primary Molars: a Randomized Clinical Trial
Brief Title: Outcomes of the Hall Technique and Conventional Pulp Therapy for the Management of Caries in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa AbdEl Moniem, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-03-16
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Deep Caries; Pulpitis - Reversible

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental group) Hall Technique (Experimental): Clinical examination to assess the clinical inclusion criteria. Radiographic examination.The child will be positioned upright in the dental chair . The correct size of PMC for the tooth will be selected. The tooth will be rinsed and dried, and the PMC dried. The PMC will be filled with glass ionomer luting cement. The PMC will be placed evenly over the tooth and the child instructed to bite down firmly until the crown was pushed down over the tooth;If the child was unable or unwilling to bite down on the PMC, finger pressure will be used to seat the crown Extruded cement will be removed, and the child will be asked to keep biting on the Hall PMC until the cement sets and once cement sets, excess cement is removed, floss will be used to clear the aproximal contacts, and post-fitting instructions will be given (Innes et al. 2007).
  Interventions: Other: Hall Technique
- Group B (control group) Formecresol Pulpotomy (Active Comparator): Clinical examination to assess the clinical inclusion criteria. Radiographic examination. The teeth anesthetized, rubber dam isolation, Complete caries removal achieved with a sterile round steel bur in a slow- speed handpiece. Access to the pulp chamber performed using a sterile slow-speed round steel bur. The pulp amputation with a sterile diamond bur in a high-speed handpiece and pulpal debris removed with a sterile saline solution on a sterile cotton pledget. After pulp amputation haemostasis achieved using a sterile cotton pledget. Formocresol (FC) applied using a sterile cotton pledget for 5 minutes. After removal of the formocresol soaked cotton pledget, the pulp chamber rinsed with water using an air-water syringe. The pulp chamber dried with a sterile cotton pledget, followed by application of Zinc Oxide & Eugenol and zinc phosphate. Tooth preparation done to receive stainless steel crown.
  Interventions: Other: Formecresol Pulpotomy

INTERVENTIONS:
Other: Hall Technique — The Hall technique is a simplified method of utilizing stainless steel crowns in treatment of carious primary molars. The SSC is cemented onto the carious tooth using glass ionomer cement. Since there is no need for carious lesion removal, the use of local anesthesia is not mandate
  Arms: Group A (Experimental group) Hall Technique
Other: Formecresol Pulpotomy — Pulpotomy is a procedure in which the coronal pulp is amputated, and the remaining radicular pulp tissue is treated with a medicament to preserve the pulp's health .This technique involves administration of local analgesia, Isolation of the tooth with rubber dam, Complete caries removal and then access to the pulp chamber using drills
  Arms: Group B (control group) Formecresol Pulpotomy

SUMMARY:
Based on the changing understanding of carious bioﬁlm development and caries progression, Sealing carious dentine beneath a restoration deprives the caries bioﬁlm of nutrients and alters the environment sufﬁciently to slow or arrest lesion progression. This has the added beneﬁt of avoiding pulp exposure and subsequent treatment .The evidence base supporting the biological approaches which include Hall technique has been steadily increasing in the last few years. This has given rise to a growing trend towards a biological approach by Paediatric dentists and has led to an increasing concern about the merits of conventional approach in treatment of carious primary molars .

DETAILED DESCRIPTION:
In orofacial development of the child, preservation of the primary dentition for as long as possible is of great importance. As primary teeth maintain arch length and preserve masticatory function. Unfortunately, the occurrence of cavitated caries lesions is still a problem in developed and developing countries, with an increasing prevalence, particulary in developing communities, conflicting with a general descending trend in prevalence worldwide.

The management of carious primary molars in children is problematic, additionally, primary teeth commonly remain unrestored, especially in the younger children,The high levels of dental disease in primary teeth, and its inadequate management, remains a major public health issue for children, and one with a significant impact on their lives. In addition many children are having to accept toothache as a part of their childhood. Set against this background, there would seem to be some scope for the investigation of alternative approaches to the management of carious primary teeth. If an alternative technique was found to be simpler and more acceptable to children, their parents and general dental practitioners than the conventional restorative approach, yet just as effective, then it might be more readily applied in the general practice setting.

A novel, simplified method of using stainless steel crwons, the Hall Technique, has been investigated. According to American Academy of Pediatric Dentistry, Hall technique calls for cementation of a Stainless steel crown over a caries-affected primary molar without local anesthetic, caries removal or tooth preparation, This technique was developed for use when delivery of ideal treatment wasn't feasible.

As the crown is fitted with no occlusal reduction in the Hall technique, it was observed in several studies that the occlusion would has been temporarily opened and returned to the pretreatment situation within 2 weeks and no child reported Tempromandibular joint pain. This goes in accordance with the study of Innes et al., as they stated that after placement of stainless steel crowns using the Hall technique, the occlusion returns to the pretreatment situation within 15-30 days. Also, Dr. Hall stated that the occlusion tended to equilibrate by the next recall appointment and none of her patients reported Tempromandibular joint pain.

A published data from Dr Hall's practice records has indicated that Hall technique might have similar survival rates to other, more conventional, restorative options currently being used in Primary Care. In addition, avoiding the use of Local anesthesia and rotary instruments for tooth preparation and caries removal might mean that the technique is less demanding of both children and their dental team. The technique is therefore minimally invasive and can be expected to cause less discomfort than conventional treatment approaches. This aspect could be a considerable advantage as the Hall technique is a child centered approach and it is not surprising that the first data published on patient perceptions of the hall technique are promising. It was reported a clear difference in levels of discomfort, subjectively assessed by the operators, between the Hall technique and a conventional treatment approach. The Hall stainless steel crowns caused 'no discomfort' to 'mild discomfort' in comparison to the conventional restorations. Several conducted studies showed that the majority of the children, their caretakers and dentists expressed a preference for the Hall technique to the conventional restorations.

The Hall Technique embraces changing concepts of managing dental caries, moving from the dogma requiring its complete surgical excision, even at the expense of cavity size and pulpal health, to the understanding that caries in dentine can be slowed, arrested, and possibly even reversed, within a meticulously sealed environment. It is known that the microflora in sealed carious dentine changes, with the predominating organisms no longer being cariogenic having been sealed from the oral environment. This may be important in the apparent arrest of caries progression.

Owing to its non invasive design, acceptance by patients and rate of restoration longevity, the Hall technique maybe an improved treatment option to increase access to care, decrease rates of untreated caries and provide a restoration that will allow for natural tooth exfoliation.

In the last few years, conventional restorations including complete removal of carious tissue with or without pulp therapy for the treatment of carious lesions in primary teeth have been challenged and a more biological approach has been suggested. This has given rise to a growing trend towards a biological approach by paediatric dentists and has led to an increasing concern about the merits of the conventional approach and whether to retain this treatment modality as the standard technique in restoring primary teeth or to adopt the biological approach as the treatment norm.

ELIGIBILITY:
Inclusion Criteria:

* Children:Aged 5 to 7 years, in good general health and medically free.The parents provided a written informed consent.
* Primary molar with deep dentin caries involving occlusal and or occluso proximal surfaces.
* Vital pulp with absence of clinical signs and symptoms of irreversible pulpitis such as spontaneous pain. Only presence of pain provoked with stimulation, such as complaints of food impaction when eating is allowed.
* Absence of clinical swelling or pus exaudate or fistula of soft or periodontal tissues.
* Absence of abnormal tooth mobility
* Absence of pain on percussion

Exclusion Criteria:

* Patients experience any signs or symptoms of pulpal or periapical pathology.
* Patients with systemic diseases requiring special dental consideration.
* Unmotivated uncooperative patients.
* Patients unable to attend follow up visits.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain reported by the patient after pulpotomy and Hall Technique | 10 days postoperatively
  Postoperative pain reported by the patient after pulpotomy and Hall Technique using visual analogue scale .Scale from 0 to 9. (Point 0): No pain ,(Points 1-3): mild pain,(Points 4-6):moderate pain, (7-9): severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa A Ibraheem, MsD, Principal Investigator — Cairo University
Locations (1):
- Hanaa A Ibraheem, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed consent form, clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after completion of the study
Access Criteria: ClinicalTrials.gov
URL: http://ClinicalTrials.gov